CLINICAL TRIAL: NCT03954249
Title: A Randomized Prospective Controlled Study Evaluating the Effectiveness of Bilateral Erector Spinae Plane Blocks in Addition to Standard Multimodal Analgesia at Reducing Opioid Consumption in Patients Undergoing Elective Mammoplasty in an Ambulatory Surgical Center
Brief Title: Evaluating the Effectiveness of Bilateral ESPB in Addition to Standard Analgesia at Reducing Opioid Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-10183
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Block
Keywords: erector spinae plane block; multimodal anesthesia
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae nerve block group (Experimental): Receive multimodal analgesia and in addition erector spinae plane block
  Interventions: Procedure: Erecto Spinae nerve block
- Multimodal Analgesia group (Active Comparator): Receive standard multimodal analgesia
  Interventions: Procedure: Multimodal Analgesia

INTERVENTIONS:
Procedure: Erecto Spinae nerve block — The ESPB is a myofascial block alternative to the paravertebral block. It is performed by injecting local anesthetic in the plane between the erector spinae muscle and the spinal transverse process. The ESPB is thought to be safer than the paravertebral block because the transverse process acts as a barrier to the pleura. It has been postulated that local anesthetic spread reaches the paravertebral space and in fact, cadaveric studies have shown dye spreading to involve the ventral and dorsal rami of spinal nerves.
  Arms: Erector Spinae nerve block group
Procedure: Multimodal Analgesia — Patients in the control group will receive standard 100mg pregabalin PO, midazolam 2mg IV, fentanyl 100mcg IV.
  Arms: Multimodal Analgesia group

SUMMARY:
Study the benefits of a Erector Spinae nerve block for pain control and decrease narcotics usage after mammoplasty in an ambulatory setting

DETAILED DESCRIPTION:
Breast surgery is among the most common procedures performed at ambulatory surgery centers. Whether for cosmetic or cancer indications, mastectomy and reduction mammoplasty are being performed under general anesthesia with standard multimodal pharmacologic analgesia. Regional anesthetic techniques have become increasingly prevalent in the management of postoperative analgesia. In oncologic surgery, regional anesthetic techniques have demonstrated a lower incidence of recurrence or metastasis of breast cancer compared to opioid analgesia. The breast has complex innervation, receiving innervation from C5-T7, thus posing a challenge to the regional anesthesiologist.

Current regional techniques for breast and other thoracic surgeries, such as open heart surgery, include the PEC I, PEC II, serratus anterior block as well as the paravertebral block. Of these options, the paravertebral block is heralded as the gold standard for multimodal analgesia in breast surgery. Unfortunately, the paravertebral block carries with it the risk of pneumothorax due to its proximity to the pleura. This risk is also increased when an inexperienced provider is performing the block, which is common on an academic institution. As a result, the PEC I, PEC II and serratus anterior blocks have gained traction, is that they carry less risk of adverse events. One drawback of the PEC blocks and serratus anterior block is that they may not achieve adequate anterior spread and complete coverage of the surgical field, making them less effective at providing adequate post-operative analgesia. Due to these drawbacks, the erector spinae plane block (ESPB) has begun to gain traction as the regional technique of choice for breast surgery. The ESPB is a myofascial block alternative to the paravertebral block. [1] It is performed by injecting local anesthetic in the plane between the erector spinae muscle and the spinal transverse process. The ESPB is thought to be safer than the paravertebral block because the transverse process acts as a barrier to the pleura. It has been postulated that local anesthetic spread reaches the paravertebral space and in fact, cadaveric studies have shown dye spreading to involve the ventral and dorsal rami of spinal nerves. It is because of this mechanism of action that this block has been call the "paravertebral by proxy." The spread of the local anesthetic is volume-dependent, and has been seen to anesthetize between 3-8 vertebral levels when using local anesthetic volumes of 15-20mL. The ESPB has been used successfully for analgesia in open-heart surgery as well as in chronic thoracic neuropathy secondary to herpetic neuralgia. Proponents of the erector spinae block prefer it to the paravertebral block for its ease to perform and seemingly safer profile.

The investigators seek to explore the proposed benefits of the erector spinae plane block in our patients undergoing bilateral breast reduction mammoplasty. Reducing overall opioid use and enhancing recovery after surgery are areas of great importance in the ambulatory, outpatient setting. The investigators hope to show the positive impact of ESPB on both of important perioperative factors.

UPDATE (1/27/2026): The 'actual' Enrollment total has been updated from 76 to 78 on account of an error identified from the time the record was completed in May 2022.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing reduction mammoplasty
* Age >18 years
* ASA class I-III

Exclusion Criteria:

* Patient refusal
* Renal insufficiency (defined as CKD stage 3 or greater)
* Infection at the skin at the site of needle puncture
* Known allergies to any study drugs
* Coagulopathy
* Severe asthmatics
* BMI >40
* ASA 4 and 5
* Pre-existing pain disorder
* Regular consumption of chronic pain medication
* Failed block
* Diagnosis of OSA

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Use of narcotics in first 24 hours | 24 hours
  The cumulative dose of oral morphine equivalence used in the 24 hours post surgery in morphine equivalents.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | Up to 1 day after surgery
  The occurrence of nausea and vomiting a subject encounters until they discharge from hospital.
Length of stay in PACU | Up to 5 Hours in PACU
  The amount of hours a subject stays in post anesthesia care unit (PACU).The time from arrival to PACU until discharge from PACU will be taken.
Assessment of postoperative pain | Up to 5 Hours in PACU
  Assessment of pain at different time points after surgery with an 11 point Numerical Rating Score(NRS) where 0 means no pain and 10 means worst imaginable pain.
Patient Satisfaction | Up to 1 day after surgery
  Assessment of patient satisfaction via a seven-point Likert scale, where 1 means extremely unsatisfied and 7 means extremely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Elilary Montilla Medrano, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No